CLINICAL TRIAL: NCT04178993
Title: A Novel Drug Combination as a Pharmacotherapeutic for Methamphetamine-Use Disorder
Brief Title: Behavioral Effects of Drugs (Inpatient): 40 [Methamphetamine, Methylphenidate, Duloxetine]
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Craig Rush (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Craig Rush, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: BED(IN):40; R01DA047391 (NIH)
Record Dates: First submitted 2019-08-09; First posted 2019-11-26 (Actual); Results first posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Methamphetamine Use Disorder
Keywords: Methamphetamine; Methylphenidate; Duloxetine Hydrochloride; Central Nervous System Stimulants; Physiological Effects of Drugs; Dopamine Uptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors; Membrane Transport Modulators; Neurotransmitter Agents; Dopamine Agents; Molecular Mechanisms of Pharmacological Action; Sensory System Agents; Peripheral Nervous System Agents; Vasoconstrictor Agents; Antidepressive Agents; Psychotropic Drugs
MeSH Terms: interventions — Methamphetamine; Methylphenidate; Lactose; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator: Placebo (Placebo Comparator): Subjects will be maintained on oral placebo. Subjects will be maintained on placebo and methylphenidate during placebo maintenance. Methamphetamine will be administered acutely during placebo maintenance. Placebo will be administered acutely during placebo maintenance.
  Interventions: Drug: Methamphetamine; Drug: Methylphenidate; Drug: Placebo oral capsule
- Active Comparator: Duloxetine (Active Comparator): Subjects will be maintained on oral duloxetine. Subjects will be maintained on duloxetine and methylphenidate during placebo maintenance. Methamphetamine will be administered acutely during duloxetine maintenance. Placebo will be administered acutely during duloxetine maintenance.
  Interventions: Drug: Methamphetamine; Drug: Methylphenidate; Drug: Placebo oral capsule; Drug: Duloxetine

INTERVENTIONS:
Drug: Methamphetamine — In each arm, subjects will receive doses of methamphetamine.
  Other Names: Metamfetamine
Drug: Methylphenidate — In each arm, subjects will receive methylphenidate capsules.
  Other Names: Metadate®
Drug: Placebo oral capsule — In each arm, subjects will receive placebo capsules.
  Other Names: Lactose
Drug: Duloxetine — Subjects will receive duloxetine capsules in the duloxetine arm.
  Other Names: Cymbalta®
  Arms: Active Comparator: Duloxetine

SUMMARY:
This study will evaluate the behavioral effects of methamphetamine during maintenance on placebo, duloxetine, methylphenidate and duloxetine combined with methylphenidate using sophisticated human laboratory methods.

ELIGIBILITY:
Inclusion Criteria:

* recent use of inhaled (i.e., snorted), smoked or injected methamphetamine

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant.
* Current or past histories of substance use that are deemed by the study physicians to interfere with study completion.
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation.
* Females not currently using effective birth control.
* Contraindications to methamphetamine, methylphenidate, or duloxetine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - University of Kentucky Medical Center, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Started | 4 | 4
Completed | 3 | 4
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38 (13.08) | 41.5 (13.11) | 39.75 (11.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 4 | 6
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Reinforcing Effects of Methamphetamine Following Methylphenidate (0 mg; Placebo) Maintenance.
Description: Number of methamphetamine doses earned by subjects on a progressive ratio schedule of reinforcement. Subjects sample a dose of methamphetamine (0, 10, or 20 mg) and then have ten opportunities (e.g., trials) to "work" for a 1/10th of the sampled dose via clicking on a computer mouse (i.e., 10 completed trials is the full sampled dose).
Time Frame: Following at least 4 days of maintenance on placebo during inpatient admission, up to 1 week
Measure: Mean (Standard Deviation); unit: Trials Completed
Groups:
- Active Comparator: Duloxetine (60 mg): Subjects will be maintained on oral duloxetine. Subjects will be maintained on duloxetine and methylphenidate during placebo maintenance. Methamphetamine will be administered acutely during duloxetine maintenance. Placebo will be administered acutely during duloxetine maintenance.
  Methamphetamine: In each arm, subjects will receive doses of methamphetamine.
  Methylphenidate: In each arm, subjects will receive methylphenidate capsules.
  Placebo oral capsule: In each arm, subjects will receive placebo capsules.
  Duloxetine: Subjects will receive duloxetine capsules in the duloxetine arm.
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine (60 mg)
Number analyzed (Participants) | 3 | 4
Trials Completed
  Methamphetamine (0mg) | 0 (0) | 0 (0)
  Methamphetamine (10mg) | 3.33 (5.77) | 7.25 (4.86)
  Methamphetamine (20mg) | 10 (0) | 9.75 (0.50)

2. Primary Outcome: Reinforcing Effects of Methamphetamine Following Methylphenidate (20 mg) Maintenance.
Description: Number of methamphetamine doses earned by subjects on a progressive ratio schedule of reinforcement. Subjects sample a dose of methamphetamine (0, 10, or 20 mg) and then have the ten opportunities (e.g., trials) to "work" for a 1/10th of the sampled dose via clicking on a computer mouse (i.e., 10 completed trials is the full sampled dose).
Time Frame: Following at least 4 days of maintenance on drug during inpatient admission, up to 1 week
Measure: Mean (Standard Deviation); unit: Trials Completed
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine (60 mg)
Number analyzed (Participants) | 3 | 4
Trials Completed
  Methamphetamine (0mg) | 0 (0) | 2.50 (5.00)
  Methamphetamine (10mg) | 6.67 (5.77) | 7.00 (4.69)
  Methamphetamine (20mg) | 8.00 (3.46) | 9.75 (0.50)

3. Primary Outcome: Reinforcing Effects of Methamphetamine Following Methylphenidate (40 mg) Maintenance.
Description: as for outcome 2
Time Frame: Following at least 4 days of maintenance on drug during inpatient admission, up to 1 week
Measure: Mean (Standard Deviation); unit: Trials Completed
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Trials Completed
  Methamphetamine (0mg) | 1.67 (2.89) | 0 (0)
  Methamphetamine (10mg) | 10 (0) | 5.00 (5.77)
  Methamphetamine (20mg) | 10 (0) | 10 (0)

4. Primary Outcome: Reinforcing Effects of Methamphetamine Following Methylphenidate (60 mg) Maintenance.
Description: as for outcome 2
Time Frame: Following at least 4 days of maintenance on drug during inpatient admission, up to 1 week
Measure: Mean (Standard Deviation); unit: Trials Completed
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine (60 mg)
Number analyzed (Participants) | 3 | 4
Trials Completed
  Methamphetamine (0mg) | 2.33 (4.04) | 0 (0)
  Methamphetamine (10mg) | 3.33 (5.77) | 7.50 (5.00)
  Methamphetamine (20mg) | 10 (0) | 9.75 (0.50)

5. Secondary Outcome: Heart Rate After Methamphetamine Administration Following Methylphenidate (0 mg) Maintenance.
Description: Heart Rate (beats per minute) is recorded following administration of methamphetamine. Data are presented as mean peak effect. Peak effect means the highest rated value following administration of methamphetamine (0, 10, and 20 mg)
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Beats Per Minute
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Beats Per Minute
  Methamphetamine (0 mg) | 77.67 (16.17) | 78.00 (6.98)
  Methamphetamine (10 mg) | 87.33 (15.14) | 77.25 (15.37)
  Methamphetamine (20 mg) | 81.33 (12.01) | 83.75 (15.20)

6. Secondary Outcome: Heart Rate After Methamphetamine Administration Following Methylphenidate (20 mg) Maintenance.
Description: as for outcome 5
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Beats Per Minute
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Beats Per Minute
  Methamphetamine (0 mg) | 83.67 (2.06) | 76.00 (8.41)
  Methamphetamine (10 mg) | 84.33 (8.50) | 78.50 (15.63)
  Methamphetamine (20 mg) | 85.67 (8.74) | 89.50 (16.90)

7. Secondary Outcome: Heart Rate After Methamphetamine Administration Following Methylphenidate (40 mg) Maintenance.
Description: as for outcome 5
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Beats Per Minute
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Beats Per Minute
  Methamphetamine (0 mg) | 85.00 (13.08) | 91.25 (23.47)
  Methamphetamine (10 mg) | 89.67 (10.21) | 87.75 (17.50)
  Methamphetamine (20 mg) | 87.67 (12.86) | 87.00 (15.08)

8. Secondary Outcome: Heart Rate After Methamphetamine Administration Following Methylphenidate (60 mg) Maintenance.
Description: as for outcome 5
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Beats Per Minute
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Beats Per Minute
  Methamphetamine (0 mg) | 87.33 (15.28) | 88.00 (19.11)
  Methamphetamine (10 mg) | 83.67 (11.72) | 87.50 (10.50)
  Methamphetamine (20 mg) | 99.67 (10.69) | 88.00 (19.36)

9. Secondary Outcome: Systolic Blood Pressure After Methamphetamine Administration Following Methylphenidate (0 mg) Maintenance.
Description: Systolic blood pressure (millimeter of mercury) is recorded following administration of methamphetamine. Data are presented as mean peak effect. Peak effect means the highest rated value following administration of methamphetamine (0, 10, and 20 mg)
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeter of Mercury
  Methamphetamine (0 mg) | 132.67 (2.89) | 128.75 (16.58)
  Methamphetamine (10 mg) | 133.00 (13.45) | 131.00 (11.83)
  Methamphetamine (20 mg) | 132.67 (5.03) | 144.25 (14.08)

10. Secondary Outcome: Systolic Blood Pressure After Methamphetamine Administration Following Methylphenidate (20 mg) Maintenance.
Description: as for outcome 9
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeter of Mercury
  Methamphetamine (0 mg) | 129.67 (2.31) | 124.25 (25.02)
  Methamphetamine (10 mg) | 131.67 (18.61) | 128.00 (17.22)
  Methamphetamine (20 mg) | 130.33 (13.20) | 132.75 (15.95)

11. Secondary Outcome: Systolic Blood Pressure After Methamphetamine Administration Following Methylphenidate (40 mg) Maintenance.
Description: as for outcome 9
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeter of Mercury
  Methamphetamine (0 mg) | 133.33 (2.08) | 129.75 (11.47)
  Methamphetamine (10 mg) | 129.00 (12.77) | 132.25 (15.41)
  Methamphetamine (20 mg) | 130.00 (10.44) | 139.25 (11.67)

12. Secondary Outcome: Systolic Blood Pressure After Methamphetamine Administration Following Methylphenidate (60 mg) Maintenance.
Description: as for outcome 9
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeter of Mercury
  Methamphetamine (0 mg) | 139.00 (4.00) | 127.00 (15.06)
  Methamphetamine (10 mg) | 138.67 (11.59) | 129.75 (14.97)
  Methamphetamine (20 mg) | 139.67 (3.06) | 135.25 (15.39)

13. Secondary Outcome: Diastolic Blood Pressure After Methamphetamine Administration Following Methylphenidate (0 mg) Maintenance.
Description: Diastolic blood pressure (millimeter of mercury) is recorded following administration of methamphetamine. Data are presented as mean peak effect. Peak effect means the highest rated value following administration of methamphetamine (0, 10, and 20 mg)
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeter of Mercury
  Methamphetamine (0 mg) | 80.00 (3.00) | 78.50 (7.77)
  Methamphetamine (10 mg) | 82.33 (0.58) | 83.75 (9.54)
  Methamphetamine (20 mg) | 87.33 (5.51) | 86.25 (7.89)

14. Secondary Outcome: Diastolic Blood Pressure After Methamphetamine Administration Following Methylphenidate (20 mg) Maintenance.
Description: as for outcome 13
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeter of Mercury
  Methamphetamine (0 mg) | 81.67 (4.51) | 74.50 (10.02)
  Methamphetamine (10 mg) | 85.33 (8.50) | 83.25 (11.03)
  Methamphetamine (20 mg) | 83.00 (3.61) | 85.00 (7.96)

15. Secondary Outcome: Diastolic Blood Pressure After Methamphetamine Administration Following Methylphenidate (40 mg) Maintenance.
Description: as for outcome 13
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeter of Mercury
  Methamphetamine (0 mg) | 78.00 (2.65) | 81.00 (9.56)
  Methamphetamine (10 mg) | 84.67 (5.51) | 82.25 (8.10)
  Methamphetamine (20 mg) | 84.67 (6.51) | 85.00 (6.06)

16. Secondary Outcome: Diastolic Blood Pressure After Methamphetamine Administration Following Methylphenidate (60 mg) Maintenance.
Description: as for outcome 13
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeter of Mercury
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeter of Mercury
  Methamphetamine (0 mg) | 82.67 (5.51) | 82.25 (5.74)
  Methamphetamine (10 mg) | 81.67 (8.08) | 82.25 (7.93)
  Methamphetamine (20 mg) | 88.33 (4.73) | 84.25 (10.37)

17. Secondary Outcome: Temperature After Methamphetamine Administration Following Methylphenidate (0 mg) Maintenance.
Description: Oral temperature (degrees fahrenheit) is recorded following administration of methamphetamine. Data are presented as mean peak effect. Peak effect means the highest rated value following administration of methamphetamine (0, 10, and 20 mg)
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Degrees Fahrenheit
  Methamphetamine (0 mg) | 98.10 (0.26) | 98.45 (0.10)
  Methamphetamine (10 mg) | 98.23 (0.40) | 98.48 (0.21)
  Methamphetamine (20 mg) | 98.40 (0.36) | 98.48 (0.19)

18. Secondary Outcome: Temperature After Methamphetamine Administration Following Methylphenidate (20 mg) Maintenance.
Description: as for outcome 17
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Degrees Fahrenheit
  Methamphetamine (0 mg) | 98.37 (0.23) | 98.50 (0.08)
  Methamphetamine (10 mg) | 98.10 (0.36) | 98.75 (0.26)
  Methamphetamine (20 mg) | 98.27 (0.32) | 98.35 (0.10)

19. Secondary Outcome: Temperature After Methamphetamine Administration Following Methylphenidate (40 mg) Maintenance.
Description: as for outcome 17
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Degrees Fahrenheit
  Methamphetamine (0 mg) | 98.17 (0.15) | 98.60 (0.22)
  Methamphetamine (10 mg) | 98.13 (0.40) | 98.65 (0.17)
  Methamphetamine (20 mg) | 98.43 (0.15) | 98.55 (0.26)

20. Secondary Outcome: Temperature After Methamphetamine Administration Following Methylphenidate (60 mg) Maintenance.
Description: as for outcome 17
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Degrees Fahrenheit
  Methamphetamine (0 mg) | 98.37 (0.35) | 98.65 (0.17)
  Methamphetamine (10 mg) | 98.43 (0.15) | 98.65 (0.06)
  Methamphetamine (20 mg) | 98.47 (0.35) | 98.58 (0.10)

21. Secondary Outcome: Subjective Effects of Methamphetamine (0 mg) Administration Following Methylphenidate (0 mg) Maintenance.
Description: Subjective effects (i.e., mood) of methamphetamine are recorded following administration. Data are presented as mean peak effect. Peak effect means the highest rated value (0 - 100 mm) following administration of methamphetamine.
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 1.33 (1.53) | 0.00 (0.00)
  Restless | 1.00 (1.73) | 0.00 (0.00)
  Nervous/Anxious | 1.00 (1.73) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 1.00 (1.73) | 0.00 (0.00)
  Talkative/Friendly | 1.00 (1.73) | 0.00 (0.00)
  Irregular/Racing Heartbeat | 1.33 (2.31) | 0.00 (0.00)
  Euphoric | 0.67 (1.15) | 0.00 (0.00)
  Shaky/Jittery | 1.33 (2.31) | 0.00 (0.00)
  Active/Alert/Energetic | 1.33 (2.31) | 1.50 (3.00)
  Will Pay For | 1.33 (2.31) | 0.25 (0.50)
  Will Take Again | 1.67 (2.89) | 1.50 (3.00)
  Performance Improved | 1.33 (2.31) | 0.00 (0.00)
  Performance Impaired | 1.00 (1.73) | 0.00 (0.00)
  Stimulated | 1.00 (1.73) | 2.25 (4.50)
  Like Drug | 1.00 (1.73) | 0.00 (0.00)
  Rush | 1.00 (1.73) | 0.25 (0.50)
  High | 0.67 (1.15) | 0.00 (0.00)
  Good Effects | 1.33 (2.31) | 0.25 (0.50)
  Bad Effects | 1.00 (1.73) | 0.00 (0.00)
  Any Effect | 1.00 (1.73) | 1.25 (2.50)

22. Secondary Outcome: Subjective Effects of Methamphetamine (10 mg) Administration Following Methylphenidate (0 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 22.33 (35.28) | 0.00 (0.00)
  Restless | 1.00 (1.73) | 1.00 (2.00)
  Nervous/Anxious | 0.67 (1.15) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 3.00 (5.20) | 0.00 (0.00)
  Talkative/Friendly | 4.33 (6.66) | 12.50 (23.04)
  Irregular/Racing Heartbeat | 0.33 (0.58) | 2.25 (4.50)
  Euphoric | 15.67 (14.29) | 18.25 (36.50)
  Shaky/Jittery | 1.00 (1.73) | 0.00 (0.00)
  Active/Alert/Energetic | 15.33 (24.83) | 25.50 (34.84)
  Will Pay For | 23.00 (38.97) | 22.25 (35.98)
  Will Take Again | 46.33 (45.06) | 23.50 (32.25)
  Performance Improved | 7.00 (9.54) | 11.50 (21.05)
  Performance Impaired | 11.33 (19.63) | 0.00 (0.00)
  Stimulated | 21.33 (36.09) | 14.25 (18.15)
  Like Drug | 33.67 (57.45) | 15.00 (15.10)
  Rush | 10.67 (18.48) | 8.25 (11.32)
  High | 9.33 (16.17) | 12.00 (14.28)
  Good Effects | 12.67 (20.21) | 13.75 (15.95)
  Bad Effects | 2.67 (4.62) | 0.00 (0.00)
  Any Effect | 12.67 (20.21) | 16.00 (19.13)

23. Secondary Outcome: Subjective Effects of Methamphetamine (20 mg) Administration Following Methylphenidate (0 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 10.33 (17.90) | 0.00 (0.00)
  Restless | 0.67 (1.15) | 0.50 (1.00)
  Nervous/Anxious | 0.67 (1.15) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 0.33 (0.58) | 0.00 (0.00)
  Talkative/Friendly | 20.00 (32.05) | 13.75 (26.84)
  Irregular/Racing Heartbeat | 1.00 (1.73) | 4.25 (7.23)
  Euphoric | 21.67 (37.53) | 16.00 (25.77)
  Shaky/Jittery | 0.67 (1.15) | 0.00 (0.00)
  Active/Alert/Energetic | 35.67 (55.72) | 27.99 (30.67)
  Will Pay For | 36.67 (55.08) | 20.50 (33.81)
  Will Take Again | 50.00 (47.70) | 25.25 (25.62)
  Performance Improved | 26.33 (37.85) | 12.00 (23.34)
  Performance Impaired | 32.67 (56.58) | 0.25 (0.50)
  Stimulated | 38.33 (53.41) | 23.50 (27.09)
  Like Drug | 37.67 (54.00) | 26.25 (27.56)
  Rush | 31.33 (54.27) | 16.00 (20.54)
  High | 36.67 (55.08) | 20.50 (22.55)
  Good Effects | 30.33 (44.77) | 23.00 (23.17)
  Bad Effects | 23.67 (40.99) | 0.25 (0.50)
  Any Effect | 38.33 (43.89) | 24.50 (24.08)

24. Secondary Outcome: Subjective Effects of Methamphetamine (0 mg) Administration Following Methylphenidate (20 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 3.00 (2.65) | 0.00 (0.00)
  Restless | 1.33 (2.31) | 1.00 (2.00)
  Nervous/Anxious | 1.67 (2.89) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 1.67 (2.08) | 0.00 (0.00)
  Talkative/Friendly | 4.00 (6.93) | 0.75 (1.50)
  Irregular/Racing Heartbeat | 1.67 (2.89) | 0.25 (0.50)
  Euphoric | 4.00 (6.93) | 0.00 (0.00)
  Shaky/Jittery | 3.00 (5.20) | 0.00 (0.00)
  Active/Alert/Energetic | 3.33 (5.77) | 0.75 (1.50)
  Will Pay For | 8.00 (13.86) | 1.00 (2.00)
  Will Take Again | 11.67 (20.21) | 1.50 (3.00)
  Performance Improved | 2.67 (4.62) | 0.75 (1.50)
  Performance Impaired | 2.33 (4.04) | 0.25 (0.50)
  Stimulated | 4.67 (8.08) | 0.25 (0.50)
  Like Drug | 7.67 (13.28) | 1.50 (3.00)
  Rush | 4.67 (8.08) | 0.00 (0.00)
  High | 4.33 (7.51) | 1.50 (3.00)
  Good Effects | 4.00 (6.93) | 1.50 (3.00)
  Bad Effects | 2.67 (4.62) | 0.00 (0.00)
  Any Effect | 3.67 (6.35) | 1.50 (3.00)

25. Secondary Outcome: Subjective Effects of Methamphetamine (10 mg) Administration Following Methylphenidate (20 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 10.67 (14.36) | 0.50 (1.00)
  Restless | 2.00 (3.46) | 0.50 (1.00)
  Nervous/Anxious | 2.00 (3.46) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 0.33 (0.58) | 0.00 (0.00)
  Talkative/Friendly | 14.67 (23.69) | 13.75 (26.18)
  Irregular/Racing Heartbeat | 0.00 (0.00) | 0.00 (0.00)
  Euphoric | 22.00 (38.11) | 13.00 (26.00)
  Shaky/Jittery | 0.67 (1.15) | 0.00 (0.00)
  Active/Alert/Energetic | 17.33 (27.43) | 16.25 (23.30)
  Will Pay For | 33.33 (57.74) | 18.50 (35.68)
  Will Take Again | 40.00 (52.74) | 21.75 (34.25)
  Performance Improved | 15.00 (23.39) | 13.00 (24.68)
  Performance Impaired | 5.67 (9.81) | 0.00 (0.00)
  Stimulated | 20.33 (32.65) | 11.75 (22.19)
  Like Drug | 35.33 (56.01) | 14.00 (24.06)
  Rush | 19.00 (32.91) | 3.00 (6.00)
  High | 21.67 (37.53) | 14.25 (21.87)
  Good Effects | 21.00 (30.35) | 9.75 (15.59)
  Bad Effects | 6.33 (10.12) | 0.25 (0.50)
  Any Effect | 16.00 (19.92) | 14.75 (18.39)

26. Secondary Outcome: Subjective Effects of Methamphetamine (20 mg) Administration Following Methylphenidate (20 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 4.33 (7.51) | 0.00 (0.00)
  Restless | 9.33 (16.17) | 1.00 (2.00)
  Nervous/Anxious | 3.33 (5.77) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 1.67 (2.89) | 0.50 (1.00)
  Talkative/Friendly | 22.67 (37.54) | 14.50 (27.01)
  Irregular/Racing Heartbeat | 3.00 (5.20) | 3.50 (5.20)
  Euphoric | 33.33 (57.74) | 14.25 (22.34)
  Shaky/Jittery | 1.33 (2.31) | 0.00 (0.00)
  Active/Alert/Energetic | 30.00 (38.97) | 24.50 (25.75)
  Will Pay For | 45.67 (50.56) | 17.25 (25.89)
  Will Take Again | 48.00 (50.12) | 24.75 (28.37)
  Performance Improved | 16.67 (23.39) | 14.50 (25.77)
  Performance Impaired | 11.33 (19.63) | 0.25 (0.50)
  Stimulated | 36.67 (55.08) | 19.75 (22.97)
  Like Drug | 47.33 (50.21) | 18.75 (23.85)
  Rush | 33.33 (57.74) | 12.75 (15.65)
  High | 33.33 (57.74) | 16.50 (18.88)
  Good Effects | 35.67 (55.73) | 14.25 (12.45)
  Bad Effects | 6.33 (10.12) | 0.00 (0.00)
  Any Effect | 36.33 (55.16) | 13.75 (12.84)

27. Secondary Outcome: Subjective Effects of Methamphetamine (0 mg) Administration Following Methylphenidate (40 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 0.00 (0.00) | 0.00 (0.00)
  Restless | 0.00 (0.00) | 0.50 (1.00)
  Nervous/Anxious | 0.00 (0.00) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 0.00 (0.00) | 0.00 (0.00)
  Talkative/Friendly | 8.00 (13.86) | 0.50 (1.00)
  Irregular/Racing Heartbeat | 0.67 (1.15) | 0.00 (0.00)
  Euphoric | 7.00 (12.12) | 0.00 (0.00)
  Shaky/Jittery | 0.67 (1.15) | 0.00 (0.00)
  Active/Alert/Energetic | 10.33 (17.90) | 0.50 (0.58)
  Will Pay For | 17.33 (30.02) | 0.75 (1.50)
  Will Take Again | 23.00 (39.84) | 1.00 (2.00)
  Performance Improved | 6.67 (11.55) | 0.00 (0.00)
  Performance Impaired | 7.67 (13.28) | 0.00 (0.00)
  Stimulated | 17.33 (30.02) | 0.50 (1.00)
  Like Drug | 16.33 (28.29) | 1.25 (2.50)
  Rush | 8.00 (13.86) | 0.00 (0.00)
  High | 10.67 (18.48) | 1.25 (2.50)
  Good Effects | 8.33 (14.43) | 1.25 (2.50)
  Bad Effects | 6.33 (10.97) | 0.00 (0.00)
  Any Effect | 7.00 (12.12) | 4.25 (5.68)

28. Secondary Outcome: Subjective Effects of Methamphetamine (10 mg) Administration Following Methylphenidate (40 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 8.67 (15.01) | 5.50 (11.00)
  Restless | 5.33 (9.24) | 1.00 (2.00)
  Nervous/Anxious | 3.00 (5.20) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 2.00 (3.46) | 0.25 (0.50)
  Talkative/Friendly | 18.67 (32.33) | 13.75 (24.86)
  Irregular/Racing Heartbeat | 2.00 (2.65) | 1.25 (2.50)
  Euphoric | 30.00 (51.96) | 9.75 (19.50)
  Shaky/Jittery | 6.33 (10.12) | 0.00 (0.00)
  Active/Alert/Energetic | 22.33 (37.82) | 20.25 (26.56)
  Will Pay For | 33.00 (54.58) | 17.00 (28.77)
  Will Take Again | 39.33 (51.60) | 17.25 (28.04)
  Performance Improved | 20.00 (33.78) | 11.25 (20.55)
  Performance Impaired | 6.00 (10.39) | 2.25 (4.50)
  Stimulated | 31.33 (51.69) | 9.50 (16.38)
  Like Drug | 33.67 (54.00) | 15.00 (24.18)
  Rush | 30.00 (51.96) | 4.50 (8.35)
  High | 30.33 (51.68) | 10.25 (15.48)
  Good Effects | 31.33 (51.68) | 9.25 (13.52)
  Bad Effects | 3.67 (6.35) | 2.50 (4.36)
  Any Effect | 30.33 (49.94) | 11.50 (12.12)

29. Secondary Outcome: Subjective Effects of Methamphetamine (20 mg) Administration Following Methylphenidate (40 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 1.33 (2.31) | 0.00 (0.00)
  Restless | 0.33 (0.58) | 1.25 (2.50)
  Nervous/Anxious | 0.00 (0.00) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 0.00 (0.00) | 0.00 (0.00)
  Talkative/Friendly | 25.33 (39.55) | 15.50 (27.01)
  Irregular/Racing Heartbeat | 2.33 (4.04) | 0.75 (1.50)
  Euphoric | 33.00 (54.58) | 14.75 (29.50)
  Shaky/Jittery | 7.00 (12.12) | 1.25 (2.50)
  Active/Alert/Energetic | 28.00 (41.68) | 24.75 (27.22)
  Will Pay For | 38.00 (54.15) | 21.25 (27.71)
  Will Take Again | 41.67 (51.81) | 23.75 (26.74)
  Performance Improved | 12.33 (20.50) | 15.00 (26.77)
  Performance Impaired | 5.33 (9.24) | 0.00 (0.00)
  Stimulated | 31.67 (48.85) | 23.25 (26.89)
  Like Drug | 34.33 (49.33) | 24.75 (26.29)
  Rush | 29.00 (49.37) | 6.75 (11.59)
  High | 28.00 (47.63) | 20.50 (22.22)
  Good Effects | 35.00 (48.545) | 22.75 (22.01)
  Bad Effects | 12.00 (10.82) | 0.00 (0.00)
  Any Effect | 33.67 (49.66) | 19.50 (20.24)

30. Secondary Outcome: Subjective Effects of Methamphetamine (0 mg) Administration Following Methylphenidate (60 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 0.00 (0.00) | 0.00 (0.00)
  Restless | 0.00 (0.00) | 0.00 (0.00)
  Nervous/Anxious | 0.00 (0.00) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 0.00 (0.00) | 0.00 (0.00)
  Talkative/Friendly | 12.33 (21.36) | 0.00 (0.00)
  Irregular/Racing Heartbeat | 0.00 (0.00) | 0.50 (1.00)
  Euphoric | 15.33 (26.56) | 0.00 (0.00)
  Shaky/Jittery | 0.00 (0.00) | 0.00 (0.00)
  Active/Alert/Energetic | 14.00 (24.25) | 0.25 (0.50)
  Will Pay For | 32.33 (50.06) | 0.00 (0.00)
  Will Take Again | 31.00 (48.59) | 3.00 (4.24)
  Performance Improved | 9.00 (15.59) | 0.00 (0.00)
  Performance Impaired | 14.33 (24.83) | 0.00 (0.00)
  Stimulated | 24.00 (41.57) | 0.00 (0.00)
  Like Drug | 29.67 (47.96) | 0.50 (1.00)
  Rush | 13.33 (23.09) | 0.00 (0.00)
  High | 12.00 (20.78) | 2.00 (2.45)
  Good Effects | 13.67 (23.67) | 0.75 (1.50)
  Bad Effects | 3.00 (5.20) | 0.00 (0.00)
  Any Effect | 15.33 (26.56) | 3.50 (5.74)

31. Secondary Outcome: Subjective Effects of Methamphetamine (10 mg) Administration Following Methylphenidate (60 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 0.00 (0.00) | 0.00 (0.00)
  Restless | 5.00 (6.24) | 1.00 (2.00)
  Nervous/Anxious | 0.00 (0.00) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 4.67 (8.08) | 0.00 (0.00)
  Talkative/Friendly | 29.00 (50.23) | 11.00 (18.74)
  Irregular/Racing Heartbeat | 0.00 (0.00) | 3.75 (3.77)
  Euphoric | 28.33 (49.07) | 11.75 (16.50)
  Shaky/Jittery | 3.67 (6.35) | 2.00 (4.00)
  Active/Alert/Energetic | 25.00 (43.30) | 23.00 (23.17)
  Will Pay For | 36.00 (54.74) | 18.00 (23.19)
  Will Take Again | 33.33 (57.74) | 23.75 (23.89)
  Performance Improved | 14.67 (25.40) | 9.50 (16.44)
  Performance Impaired | 5.33 (9.24) | 0.00 (0.00)
  Stimulated | 33.00 (52.83) | 17.25 (18.19)
  Like Drug | 32.67 (55.72) | 23.75 (23.30)
  Rush | 27.33 (47.34) | 10.75 (21.50)
  High | 27.00 (46.77) | 15.75 (16.58)
  Good Effects | 25.33 (43.88) | 20.25 (18.37)
  Bad Effects | 4.67 (8.08) | 0.00 (0.00)
  Any Effect | 24.67 (41.86) | 20.75 (18.39)

32. Secondary Outcome: Subjective Effects of Methamphetamine (20 mg) Administration Following Methylphenidate (60 mg) Maintenance.
Description: as for outcome 21
Time Frame: Daily over approximately 1 week of inpatient stay.
Measure: Mean (Standard Deviation); unit: Millimeters
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine
Number analyzed (Participants) | 3 | 4
Millimeters
  Sluggish/Fatigued/Lazy | 6.67 (11.55) | 0.00 (0.00)
  Restless | 0.00 (0.00) | 1.25 (1.89)
  Nervous/Anxious | 0.33 (0.58) | 0.00 (0.00)
  Nauseated/Queasy/Sick to Stomach | 0.00 (0.00) | 0.00 (0.00)
  Talkative/Friendly | 29.33 (50.23) | 18.25 (31.94)
  Irregular/Racing Heartbeat | 30.67 (53.12) | 1.00 (2.00)
  Euphoric | 32.33 (56.00) | 18.00 (35.34)
  Shaky/Jittery | 2.00 (3.46) | 0.25 (0.50)
  Active/Alert/Energetic | 37.33 (53.46) | 21.50 (29.92)
  Will Pay For | 34.00 (57.17) | 18.75 (32.31)
  Will Take Again | 37.67 (54.04) | 21.50 (30.49)
  Performance Improved | 22.00 (33.05) | 18.75 (33.00)
  Performance Impaired | 10.33 (17.90) | 13.50 (27.00)
  Stimulated | 36.00 (53.73) | 20.25 (32.57)
  Like Drug | 36.33 (54.31) | 21.50 (31.72)
  Rush | 35.67 (53.35) | 2.50 (5.00)
  High | 37.00 (54.03) | 20.25 (27.89)
  Good Effects | 39.00 (53.23) | 20.25 (27.93)
  Bad Effects | 9.67 (16.74) | 0.00 (0.00)
  Any Effect | 38.00 (53.11) | 19.25 (24.78)

33. Other Pre Specified Outcome: Attentional Bias
Description: Subjects will complete an attentional bias task. The number of inhibitory failures (i.e., commission errors) to "no-go" targets following methamphetamine-related stimuli will be used to evaluate attentional bias (range 0 - 1: greater values represent greater number of errors committed). Commission errors are when you response (i.e., press the corresponding key on a computer) when you were instructed not to respond.
Time Frame: 12 sessions over approximately 4.5 weeks
Measure: Mean (Standard Deviation); unit: Proportion of Responses
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine (60 mg)
Number analyzed (Participants) | 3 | 4
Proportion of Responses
  Methylphenidate (0mg) | 0.07 (0.08) | 0.08 (0.07)
  Methylphenidate (20mg) | 0.04 (0.04) | 0.13 (0.09)
  Methylphenidate (40mg) | 0.08 (0.04) | 0.11 (0.05)
  Methylphenidate (60mg) | 0.12 (0.11) | 0.12 (0.06)

34. Other Pre Specified Outcome: Snaith-Hamilton-Pleasure Scale to Measure Anhedonia (Inability to Experience Pleasure)
Description: A 14-item Snaith-Hamilton-Pleasure Scale covers four domains of pleasure response (interest/pastimes, social interaction, sensory experience and food/drink) with higher scores representing less anhedonia. Scores range from 0 to 56 units: lower scores representing greater anhedonia.
Time Frame: 4 times over approximately 4.5 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine (60 mg)
Number analyzed (Participants) | 3 | 4
Units on a Scale
  Methylphenidate (0 mg) | 44.33 (8.33) | 51.25 (6.60)
  Methylphenidate (20 mg) | 44.00 (3.46) | 52.75 (4.72)
  Methylphenidate (40 mg) | 44.33 (5.51) | 54.00 (2.45)
  Methylphenidate (60 mg) | 44.67 (5.88) | 53.00 (6.00)

35. Other Pre Specified Outcome: Delay Discounting for Methamphetamine
Description: Subjects will complete a delay discounting task in 4 sessions following 4 days of medication maintenance. Subjects are presented a series of hypothetical choices between a smaller amount of methamphetamine offered "now" or a larger amount of methamphetamine offered a later times in the future (e.g., 4 hours, a day, 3 weeks). The discounting rate, 'k', is calculated and log10-transformed. Greater values of log-transformed 'k' correspond with greater rates of discounting (i.e., preference for smaller reinforcer provided now rather than larger, delayed reinforcers [e.g., smaller amount of methamphetamine given now as opposed to a larger amount given later]). The units for discounting rates are theoretical and not linked to a physical dimension (e.g., number of button presses) and the range is theoretically not bound (i.e., negative infinity to positive infinity).
Time Frame: 4 sessions over approximately 4.5 weeks
Measure: Mean (Standard Deviation); unit: log(k)
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine (60 mg)
Number analyzed (Participants) | 3 | 4
log(k)
  Methylphenidate (0mg) | -1.40 (1.63) | -1.31 (0.72)
  Methylphenidate (20mg) | -1.04 (1.10) | -1.27 (0.49)
  Methylphenidate (40mg) | -1.45 (1.63) | -1.15 (0.33)
  Methylphenidate (60mg) | -1.17 (1.91) | -1.04 (0.43)

36. Other Pre Specified Outcome: Delay Discounting for Money
Description: Subjects will complete a delay discounting task in 4 sessions following 4 days of medication maintenance. Subjects are presented a series of hypothetical choices between a smaller sum of money offered "now" or a larger sum of money offered a later times in the future (e.g., 4 hours, a day, 3 weeks). The discounting rate, 'k', is calculated and log10-transformed. Greater values of log-transformed 'k' correspond with greater rates of discounting (i.e., preference for smaller reinforcer provided now rather than larger, delayed reinforcers [e.g., smaller sum of money given now as opposed to a larger sum given later]). The units for discounting rates are theoretical and not linked to a physical dimension (e.g., number of button presses) and the range is theoretically not bound (i.e., negative infinity to positive infinity).
Time Frame: 4 sessions over approximately 4.5 weeks
Measure: Mean (Standard Deviation); unit: log(k)
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine (60 mg)
Number analyzed (Participants) | 3 | 4
log(k)
  Methylphenidate (0mg) | -1.40 (1.63) | -1.29 (0.76)
  Methylphenidate (20mg) | -1.40 (1.63) | -1.37 (0.58)
  Methylphenidate (40mg) | -1.45 (1.63) | -1.15 (0.33)
  Methylphenidate (60mg) | -1.48 (1.43) | -1.04 (0.43)

ADVERSE EVENTS:
Time Frame: Assessed during 4.5 weeks of inpatient study.
Arm/Group | Placebo Comparator: Placebo | Active Comparator: Duloxetine (60 mg)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 0.29% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator: Placebo (N=3) | Active Comparator: Duloxetine (60 mg) (N=4)
Elevated Heart Rate (Cardiac disorders) | 2 (2) | 2 (2)
Elevated Blood Pressure (Cardiac disorders) | 2 (2) | 2 (2)
Migraine (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/93/NCT04178993/Prot_SAP_ICF_001.pdf